CLINICAL TRIAL: NCT05233540
Title: Circulating Biomarkers in Patients With Anal Cancer Treated With Induction Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Karen Wind, Medical Doctor, principal investigator, Aarhus University Hospital
Other Study IDs: DACG-III
Record Dates: First submitted 2022-01-25; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Anal Cancer; Locally Advanced Squamous Cell Carcinoma; Oligometastatic Disease; Circulating Tumor Cell; Human Papilloma Virus
MeSH Terms: conditions — Anus Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and diagnostic biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Locally advanced or synchronous metastatic anal cancer treated with induction chemotherapy: Patients with newly diagnosed anal cancer who by standard of care are eligible for induction chemotherapy prior to definitive CRT or radiotherapy alone (RT) will be screened according to inclusion- and exclusion criteria. Patients eligible for induction chemotherapy will be patients with locally advanced or synchronous metastatic anal cancer.

SUMMARY:
To investigate the prognostic and predictive value of plasma HPV (pHPV) prior, during and after induction chemotherapy (ICT) in locally advanced squamous cell carcinoma of the anus (SCCA) or synchronous metastatic SCCA patients treated with ICT prior to definitive (chemo)radiotherapy ((C)RT) according to multidisciplinary team (MDT) conferences based decisions. Further to investigate the use of pHPV measurements and other relevant markers for prediction of response and survival after ICT prior to definitive (C)RT.

DETAILED DESCRIPTION:
Anal cancer is a rare malignancy with approximately 200 new cases in Denmark per year, and the standard treatment is chemoradiotherapy (CRT). The treatment is centralised at three oncological departments at Aarhus University Hospital, Herlev Hospital and Vejle Hospital. The majority of anal cancers are squamous cell carcinomas (SCCA) and are strongly associated with human papilloma virus (HPV) which can be detected in tumour tissue in more than 80% of cases. Patients with large tumours, tumours invading nearby organs and/or local lymph node metastases could be treated with induction chemotherapy (ICT) in cases where downsizing prior definitive treatment is needed. Selected patients with metastatic (M1) SCCA could also be treated with ICT with the purpose of making definitive treatment possible.

HPV, cell-free DNA, circulating tumour DNA and immune related markers:

HPV is a virus group consisting of more than 130 subtypes, of which a minor part is categorised as oncogenic types. The most common HPV subtypes found in SCCA is HPV-16 and -18, but the total landscape of HPV subtype distribution in SCCA is sparsely investigated. Small fragments of cell-free DNA (cfDNA) can be detected in the circulation with elevated levels in cancer patients, but also in other circumstances. Aberrant methylation of DNA occurs in almost all malignant tumours and is shed into the circulation. The level of tumour specific methylated DNA (meth-ctDNA) can be analysed by modern PCR technology. It seems to hold biological information, which holds promise of clinical utility. The literature has focused on colorectal cancer and meth-ctDNA has been introduced as a prognostic marker. The possible importance in anal cancer has not been elucidated which is one the aims of the present protocol. With a simple blood test (so called "liquid biopsy"), it is possibility to characterise both the level of total cfDNA and meth-ctDNA. HPV associated anal cancer has a viral sequence integrated into the genome of the cancer cells. In HPV associated anal cancer meth-ctDNA is shredded to the blood stream, and can be measured as HPV tumour cell DNA (plasma HPV or pHPV). The observational and translation part of the DACG Plan-A study have shown that levels of pre-treatment pHPV are higher in large tumours compared to small and higher in node positive disease compared to node negative which is in agreement with results on advanced anal cancer where pHPV levels were correlated to tumour burden. The Plan-A study have also shown that pHPV is eliminated during CRT in case of response to treatment.

Immunotherapy has changed the treatment of several malignant tumours, especially malignant melanoma. The checkpoint inhibitors block PD/PD-L1 interaction, which elicits immune response to the malignant tumour. The treatment also seems to have effect in anal cancer. The literature is sparse, but a number of studies are ongoing. It is therefore well motivated to analyse one of the central stakeholders in the immune response. The level of PD-L1 in serum holds potential as a prognostic marker in anal cancer.

Perspective:

In patients treated with ICT prior to definitive CRT it is crucial not to exceed the necessary amount of potentially toxic treatment cycles and the ability of pHPV to address early response or progression is highly relevant. Complete response after ICT have been reported and treatment with ICT consisting of e.g. cisplatin, 5-flourouracil, leuroverin and ifosfamide (CILF) have shown a complete local tumour response rate of 15% and prediction of response is therefore highly relevant. In the metastatic setting taxol and carboplatin has now been introduced as first line option. This combination is also a relevant candidate for ICT. The potential perspective will be development of studies with pHPV guided intensified ICT.

Purpose:

To investigate the prognostic and predictive value of pHPV prior, during and after ICT in patients treated with ICT according to multidisciplinary team (MDT) conferences based decisions. Further to investigate the use of pHPV measurements and other relevant markers for prediction of response and survival after ICT prior to definitive CRT.

ELIGIBILITY:
Inclusion Criteria:

* Histological verified squamous cell carcinoma of the anus
* Treatment with ICT prior to definitive CRT or RT due to locally advanced disease or
* Patients with synchronous metastatic disease treated with ICT with the purpose of definitive CRT (potentially in combination with organ directed therapy (surgery, RFA, SBRT) for the metastatic sites)
* Age ≥ 18 years
* Written and orally informed consent

Exclusion Criteria:

* Contraindications for blood sampling
* Other malignancy within the past five years, with exception of basal cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed anal cancer who by standard of care are eligible for ICT prior to definitive CRT or radiotherapy alone (RT) will be screened according to inclusion- and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival according to circulating tumour DNA status | 2 year
  Overall survival: Time from diagnosis to time of dead or date of last follow-up.

SECONDARY OUTCOMES:
Disease-free survival according to circulating tumour DNA and immune markers. | 2 year
  Time from end of treatment to progression, recurrence or death whatever comes first.
Recurrence-free survival according to circulating tumour DNA and immune markers. | 2 year
  Time from end of treatment to recurrence (locoregional or distant failure) or death whatever comes first.
Overall survival according to circulating tumour DNA and immune markers. | 2 year
  Overall survival: Time from diagnosis to time of death or date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Wind, MD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Department of Oncology, Aarhus University Hospital, Aarhus, Aarhus N
  - Department of Oncology Herlev and Gentofte Hospital, Herlev
  - Department of Oncology, Vejle hospital, University Hospital of Southern Denmark, Vejle

IPD SHARING:
Plan to Share IPD: No